CLINICAL TRIAL: NCT00190268
Title: Multicentric Study, Comparative, Randomized, in Double Knowledge of the Effectiveness (Versus Placebo) of a Salt Of 3,4 - Diaminopyridine in the Treatment of Tiredness During the Multiple Sclerosis
Brief Title: Efficacy of 3,4-DAP in Fatigue Associated With Multiple Sclerosis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Isabelle BRINDEL, Department of Clinical Research of developpement
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: P020304; NCT00169429 (obsolete NCT alias)
Record Dates: First submitted 2005-09-13; First posted 2005-09-19 (Estimated); Last update posted 2011-02-21 (Estimated); Status verified 2007-03

CONDITIONS: Multiple Sclerosis
Keywords: multiple sclerosis; fatigue; 3,4-diaminopyridine
MeSH Terms: conditions — Multiple Sclerosis; Fatigue | interventions — Amifampridine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 3,4-diaminopyridine (Experimental): 3,4-diaminopyridine
  Interventions: Drug: 3,4-diaminopyridine

INTERVENTIONS:
Drug: 3,4-diaminopyridine — 3,4-diaminopyridine

SUMMARY:
Rational of study : 3,4-diaminopyridine is suspected to improved the fatigue associated in patient's multiple sclerosis.

In order to confirm this hypothesis, a randomized, controlled versus placebo, double blinded study is performed.

DETAILED DESCRIPTION:
We proposed a randomized controlled trial between 3,4-diaminopyridine and placebo .

The main objective : improvement of fatigue by diminution of EMIF-SEP score between the arm treatment and placebo arm. The hypothesis tested is that the 3,4-DAP is efficacy in the fatigue of multiple sclerosis.

ELIGIBILITY:
Inclusion Criteria:

* Age >= 18 years and = <60 years
* Patients with multiple sclerosis clinically defined and with MIFS-SEP score > 44, without deficit sleep and without depression.
* Patients without treatment by 3,4-DAP since 3 months
* EDSS score < 6

Exclusion Criteria:

* ASAT/ALAT > 2 x ULN
* MADRS >= 20
* Abnormality cardiac rhythm
* Pregnancy
* Asthma
* Evolutive affection
* Renal failure

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 126 (Actual)
Dates: Start 2005-02; Primary Completion 2008-06 (Actual); Study Completion 2008-06 (Actual)

PRIMARY OUTCOMES:
improvement of fatigue measured by a decrease of EMIF-SEP score compared to placebo group. | 43 months
  improvement of fatigue measured by a decrease of EMIF-SEP score compared to placebo group.

SECONDARY OUTCOMES:
evaluation of safety | 43 months
  evaluation of safety
quality of life impact | 43 months
  quality of life impact

CONTACTS AND LOCATIONS:
Overall Officials: Pierre Cesaro, MD, Study Chair — Hopital Henri Mondor-France
Locations (4):
- France (4):
  - Henri Mondor Hospital, Créteil
  - Pitié Salpetriere Hospital, Paris
  - Tenon Hospital, Paris
  - Pontchaillou Hospital, Rennes